CLINICAL TRIAL: NCT01667835
Title: Yoga for Post-menopausal South Asian Women at Risk for Cardiovascular Disease: A Randomized Control Pilot Study
Brief Title: South Asian Women & Yoga Education Study
Acronym: SAWYES
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kwantlen Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Amandah Hoogbruin, Principal Investigator, Community & Health Studies Faculty member, Kwantlen Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KK11-04
Record Dates: First submitted 2012-06-17; First posted 2012-08-17 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Cardiovascular Disease
Keywords: yoga; postmenopausal, sedentary South Asian women
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Intervention (Experimental)
  Interventions: Behavioral: Yoga Intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Yoga Intervention — 12 week 90 minute hatha yoga session offered three (3x) per week. Hatha yoga is a form of structured physical exercises known as asanas, combined with breathing exercises called pranayama, and relaxation techniques. The yoga intervention consists of 9 different yoga poses (asanas) and 3 different breathing exercises (pranayama) that can be easily replicated and readily performed by individuals who are middle-aged and older, overweight, unfit, or who suffer from a chronic illness.
  Arms: Yoga Intervention

SUMMARY:
The purpose of this randomized, control pilot study is to measure the effects of a gentle, 12 week hatha yoga program on post-menopausal, obese, sedentary South Asian women at risk for cardiovascular disease. Hatha yoga is a form of structured physical exercises known as asanas, combined with breathing exercises called pranayama, and relaxation techniques. The yoga intervention consists of 9 different yoga poses (asanas) and 3 different breathing exercises (pranayama) that can be easily replicated and readily performed by individuals who are middle-aged and older, overweight, unfit, or who suffer from a chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* 40- 65 years old
* Postmenopausal (amenorrhea for ≥ 12 months)
* Overweight as evidenced by a body mass index (BMI) ≥ 25 kg/m2), or waist circumference ≥ 80 cm, or have a first degree relative with diabetes or essential hypertension
* Sedentary, do not do a regular exercise program (exercising for 20 minutes at sufficient intensity to produce sweating less than 2x/week)
* Self-identify as a South Asian (sometimes referred to as East Indian in Canada and may be defined "as any person who reports an ethnicity associated with the southern part of Asia or who self-identifies as part of the South Asian visible minority group. This definition encompasses people from a great diversity of ethnic backgrounds, including those with Bangladeshi, Bengali, East Indian, Goan, Gujarati, Hindu, Ismaili, Kashmiri, Nepali, Pakistani, Punjabi, Sikh, Sinhalese, South Asian, Sri Lankan and Tamil ancestry. South Asians may have been born in Canada, on the Indian sub-continent, in the Caribbean, in Africa, in Great Britain or elsewhere
* Given consent to research protocol and willingness to be randomized to either the treatment (yoga) or control (no yoga) group.

Exclusion Criteria:

* Have had a period within the last year
* Are not between the ages of 40 and 65
* Have experience with yoga within the last 12 months
* Have any serious disease or condition such as diabetes, serious high blood pressure or heart problems, kidney disease, severe asthma, cancer (except for skin cancer that is not melanoma)
* Have a major brain or nervous system diagnosis, such as Parkinson's disease or stroke
* Have a severe infectious or other medical illness right now such as pneumonia
* Use medications to lower blood sugar levels
* Have serious back, hip, or neck problems or pain in joints or bones that would prevent the safe completion of a gentle 12 week Hatha yoga program
* Regularly use an assistive device (e.g., cane, walker) to walk

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-12 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | baseline, at end of study (12 wks), & 3 months post-study
  blood pressure is measured as a specific physiologic index of cardiovascular risk.

SECONDARY OUTCOMES:
Change in subjective well-being | baseline, at end of study (12 wks), & 3 months post-study
  The Perceived Stress Scale and Abbreviated Duke Social Support Index will be used to measure subjective well-being.
Change in perceived physical well-being | baseline, end of study (12 wks) & 3 months post-study
  Pittsburgh Sleep Quality Index, Physical Activity Scale for the Elderly, and Exercise Regularly Scale will be used to measure change in perceived physical well-being
Change in insulin sensitivity | baseline, end of study (12 wks) & 3 months post-study
  Fasting insulin & glucose will be measured for change in insulin sensitivity as a related index of cardiovascular risk
Change in inflammation | baseline, end of study (12 wks) & 3 months post-study
  C-reactive protein will be measured for change in inflammation as a related index of cardiovascular risk
Change in serum total cholesterol | baseline, end of study (12 wks) & 3 months post-study
  Serum total cholesterol will be measured as a related index of cardiovascular risk
Change in serum high-density lipoprotein (HDL) cholesterol | baseline, end of study (12 wks) & 3 months post-study
  Serum high-density lipoprotein (HDL) cholesterol will be measured as a related index of cardiovascular risk
Change in serum low-density lipoprotein (LDL) cholesterol | baseline, end of study (12 wks) & 3 months post-study
  Serum low-density lipoprotein (LDL)cholesterol will be measured as a related index of cardiovascular risk
Change in serum triglycerides | baseline, end of study (12 wks) & 3 months post-study
  Serum triglycerides will be measured as a related index of cardiovascular risk
Change in waist circumference. | baseline, end of study (12 wks) & 3 months post-study
  Waist circumference will be measured for change in visceral adiposity as a related index of cardiovascular risk
Change waist-hip ratio | baseline, end of study (12 wks) & 3 months post-study
  Waist-hip ratio will be measured for change in visceral adiposity as a related index of cardiovascular risk
Change in body mass index (BMI) | baseline, end of study (12 wks) & 3 months post-study
  Body mass index (BMI) will be measured for change in visceral adiposity as a related index of cardiovascular risk
Change in resting heart rate | baseline, end of study (12 wks) & 3 months post-study
  Resting heart rate will be measured for change in sympathetic activity as a related index of cardiovascular risk
Change in heart rate | baseline, at end of study (12 wks), & 3 months post-study
  Heart rate will be measured for change in sympathetic activity as a related index of cardiovascular risk

CONTACTS AND LOCATIONS:
Overall Officials: Amandah L Hoogbruin, PhD, Principal Investigator — Kwantlen Polytechnic University
Locations (2):
- Canada (2):
  - The Jim Pattison Outpatient Care and Surgery Services, Cardiovascular Outpatient Clinic, Surrey, British Columbia
  - Kwantlen Polytechnic University, Surrey, British Columbia